CLINICAL TRIAL: NCT07344311
Title: First Time-in-Human (FTiH), Phase I Trial to Evaluate the Safety, Cellular Kinetics, and Efficacy of A-CAR032, in Adult Participants With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: A Phase I Trial of A-CAR032 in Participants With mCRPC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1332-046
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Metastatic Castration-Resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A-CAR032 (Experimental): Part 1 will follow an i3+3 design which is employed to explore the maximum tolerated dose (MTD) and/or the recommended dose for expansion (RDE). Three dose levels of A-CAR032are initially planned with a minimum of 3 and maximum of 9 participants per dose level. The safety review committee (SRC) may suggest exploration of intermediate dose levels or additional higher or lower dose levels based on the available data, but will not exceed 3 times the current dose or 3 times the highest dose that has been determined safe by the SRC.Part 2 at the RDE of A-CAR032 will be initiated, if data support, to further evaluate the safety, CK, efficacy and potential biological activity of study intervention. Approximately 12 evaluable participants will be enrolled in Part 2.
  Interventions: Biological: dnTGFβRII-armoured STEAP2-targeted autologous CAR T-Cell Injection

INTERVENTIONS:
Biological: dnTGFβRII-armoured STEAP2-targeted autologous CAR T-Cell Injection — dnTGFβRII-armoured STEAP2-targeted autologous CAR T-Cell Injection.single infusion intravenously.

SUMMARY:
This FTiH, single-arm, open-label, investigator-initiated Phase I trial will evaluate the safety, antitumour activity, CK/pharmacodynamics (PD), biomarkers, immunogenicity, and feasibility of A-CAR032 in adult participants with mCRPC, who have previously progressed after ARPI treatment of prostate cancer (whether before or in the metastatic castration-resistant setting) and, in the judgment of the investigator, are ineligible for standard treatment.

DETAILED DESCRIPTION:
The study consists of two parts: Part 1-Dose Escalation and Part 2-Dose Expansion. Participants in the study will proceed through screening, apheresis, bridging therapy (if appropriate), lymphodepletion, CAR-T cell infusion, and subsequent follow-up (including Stage 1, 2 and 3).

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 years or older at the time of signing the ICF. Type of Participant and Disease Characteristics
2. Participants with:

   1. A histologically confirmed diagnosis of metastatic adenocarcinoma of the prostate without known neuroendocrine differentiation or small cell features.
   2. Castration-resistant prostate cancer as defined by disease progression despite castration by orchiectomy or ongoing luteinising hormone-releasing hormone analogue. Participants receiving medical castration therapy with gonadotropin-releasing hormone analogues should continue this treatment during the study.
   3. Measurable PSA≥1 ng/mL AND
   4. Evidence of progression within 6 months prior to screening
3. Participant has previously received an ARPI (ie, abiraterone, enzalutamide, apalutamide, darolutamide, rezvilutamide) whether before or in the metastatic castration-resistant setting, and in the judgment of the investigator, be ineligible for standard treatment.
4. Minimum life expectancy of > 12 weeks prior to apheresis in the opinion of the investigator.
5. Adequate organ and marrow function
6. Consent and provision of tumour material to assess STEAP2 expression and other correlative biomarkers retrospectively with pre- and post-treatment biopsies.
7. Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
8. The participant voluntarily participates in the study, and the individual or their legal guardian signs the ICF.

Exclusion Criteria:

1. Known life-threatening allergies, hypersensitivity, or intolerance to the CAR-T product or its excipients, including dimethyl sulfoxide (DMSO).
2. Contraindication to lymphodepleting agents, including fludarabine and/or cyclophosphamide.
3. History of another primary malignancy except for:

   1. Malignancy treated with curative intent and with no known active disease within 3 years before the apheresis and of low potential risk for recurrence.
   2. Adequately treated non-melanoma skin cancer or lentigo malignancy without evidence of disease.
   3. Adequately treated carcinoma in situ without evidence of disease.
4. Participants with known brain metastases.
5. History of splenectomy or organ transplantation.
6. Prior treatment with:

   1. Any CAR-T therapy. OR
   2. Any therapy that is targeting STEAP2.
7. Active or prior documented autoimmune or inflammatory disorders
8. Cardiac arrhythmias which are symptomatic or require treatment unless controlled by pacemaker (judged by investigator); symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia.
9. Active infection, including:

   1. HBV infection is defined as hepatitis B surface antigen (HBsAg) positive, or hepatitis B core antibody (HBcAb) positive and HBV DNA detectable.
   2. HCV infection is defined as HCV antibody positive and HCV RNA positive.
   3. CMV infection is defined as CMV DNA detectable.
   4. Syphilis infection is defined as syphilis antigen and antibody positive.
   5. HIV infection is defined as HIV 1/2 antibody positive.
   6. Other persistent or active infections requiring systemic treatment (prophylactic use of anti-infective drugs is allowed).
10. Patients with central nervous system (CNS) diseases:
11. Obvious risk or tendency of bleeding or active bleeding (eg, clinically significant hemoptysis, tumour bleeding, history of von Willebrand disease or hemophilia etc.).
12. Plans to father a child during the study period.
13. Patients with alcohol or drug abuse.
14. Participants may not receive full-dose long acting oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose from the time of informed consent to 28 days post infusion of A-CAR032. Use of short acting direct oral anticoagulants for therapeutic and prophylactic purposes are permitted.
15. Received the following:

    1. Major surgery within 4 weeks prior to apheresis or existence of unhealed wound, or planned major surgery within 4 weeks of the study treatment administration
    2. Steroids (except inhaled steroids) or other immunomodulators (including interleukins, interferons, and thymosins) of systemic therapeutic dose, and systemic corticosteroids at doses exceeding 10 mg/day of prednisone or equivalent within 5 half-lives or 7 days (whichever is shorter) prior to apheresis.
16. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy targeted therapy, biologic therapy, tumour embolisation, or monoclonal antibodies, investigational product) within 5 half-lives or ≤ 21 days (whichever is shorter) prior to apheresis.
17. Radiotherapy within 4 weeks of apheresis (However, if the radiation portal covered ≤ 5% of the bone marrow reserve, the participant is eligible irrespective of the end date of radiotherapy); or within 6 months or 5 half-lives (whichever is longer) if local radioactive particle implantation was performed.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2042-01-31 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation (Part 1)：Safety | From ICF signature until 15 years post A-CAR032 infusion
  Incidence of AEs/SAEs
Dose Escalation (Part 1)：Safety | Throughout the 28 days post A-CAR032 infusion
  Occurrence of DLTs/DLT-like events
Dose Escalation (Part 1)：Safety | From ICF signature until 12 months post A-CAR032 infusion
  Changes from baseline in laboratory parameters, vital signs, and ECGs
Dose Expansion (Part 2)：Safety | From ICF signature until 15 years post A-CAR032 infusion
  Incidence of AEs/SAEs
Dose Expansion (Part 2)：Safety | Throughout the 28 days post A-CAR032 infusion
  Incidence of DLT-like events
Dose Expansion (Part 2)：Safety | From ICF signature until 12 months post A-CAR032 infusion
  Changes from baseline in laboratory parameters, vital signs, and ECGs

SECONDARY OUTCOMES:
Dose Escalation (Part 1) and Dose Expansion (Part 2)：Efficacy | From ICF signature until 12 months post A-CAR032 infusion
  PSA-related response
Dose Escalation (Part 1) and Dose Expansion (Part 2)：Efficacy | From ICF signature until 12 months post A-CAR032 infusion
  Radiological response
Dose Escalation (Part 1) and Dose Expansion (Part 2)：Efficacy | From ICF signature until 12 months post A-CAR032 infusion
  rPFS
Dose Escalation (Part 1) and Dose Expansion (Part 2)：Efficacy | From ICF signature until 15 years post A-CAR032 infusion
  OS
Dose Escalation (Part 1) and Dose Expansion (Part 2)：Efficacy | From A-CAR032 infusion until 12 months post A-CAR032 infusion
  Time from A-CAR032 infusion to first SSRE
Dose Escalation (Part 1) and Dose Expansion (Part 2)：Pharmacokinetics | From ICF signature until 15 years post A-CAR032 infusion
  CK profile of A-CAR032

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No